CLINICAL TRIAL: NCT06711991
Title: A Phase I Clinical Study on the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Characteristics of Single/Multiple Dose Escalation of TQC3927 Inhalation Powder in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Clinical Trial of TQC3927 Powder for Inhalation in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC3927-I-02
Record Dates: First submitted 2024-11-22; First posted 2024-12-02 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC3927 powder for inhalation (Experimental): TQC3927 powder for inhalation is administered as a single administration for 1 day and continuous administration for 6 days.
  Interventions: Drug: TQC3927 powder for inhalation
- TQC3927 powder for inhalation placebo (Active Comparator): TQC3927 powder for inhalation placebo is administered as a single administration for 1 day and continuous administration for 6 days.
  Interventions: Drug: TQC3927 powder for inhalation placebo

INTERVENTIONS:
Drug: TQC3927 powder for inhalation — TQC3927 is a targeted inhibitor
  Arms: TQC3927 powder for inhalation
Drug: TQC3927 powder for inhalation placebo — A placebo without drug substance.
  Arms: TQC3927 powder for inhalation placebo

SUMMARY:
This project is the stage of dose escalation, is was divided into single and multiple dose clinical study, This is a multi-center, randomized, double-blind, placebo-controlled , study to the safety, tolerability and pharmacokinetic characteristics of TQC3927 powder for inhalation in Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years (inclusive)，both male and female
* The subjects were able to undergo reproducible FEV1 lung function testing according to the American Thoracic Society/European Respiratory Society (ATS/ERS) 2005 standard during screening
* Subject should weigh at least 45kg. And body mass index (BMI) within 18~30 kg/m2
* Have no pregnancy plan and voluntarily take effective contraception measures from time of screening to at least 90 days after the last dose (subjects and their partners)

Exclusion Criteria:

* Patients with a history of glaucoma, functional constipation, prostate hyperplasia, urinary tract obstruction, etc
* Individuals with a history of illegal drug abuse or who have tested positive for drug abuse screening during the screening period (including benzodiazepines, methamphetamine, cocaine, morphine, ketamine, tetrahydrocannabinol)
* Participated in other clinical trials and received research interventions in the 3 months prior to participating in this trial
* Screening for individuals who have used biologics within the past 3 months
* Individuals who have lost blood or donated more than 400 mL of blood within 3 months prior to the experiment, or who have received blood transfusions or used blood products
* Any clear history of drug or food allergies, especially those who are allergic to ingredients similar to the investigational drug
* Screening for individuals who have frequently consumed alcohol within the previous 6 months (i.e. females consume more than 14 standard units of alcohol per week, males consume more than 21 standard units of alcohol per week (1 standard unit contains 14g of alcohol, such as 360 mL beer or 45 mL of 40% alcohol strong liquor or 150 mL wine) or are unable to abstain from alcohol during the trial period; Or those who test positive for alcohol breath test
* History of any malignant tumors in organs or systems within the past 5 years, regardless of whether they have received treatment or not, except for local basal cell carcinoma of the skin
* When screening, the sitting systolic blood pressure should be ≥ 160 mmHg, and the sitting diastolic blood pressure should be ≥ 100 mmHg; Pulse rate<50 bpm or>100 bpm
* Clinically significant apnea patients requiring continuous positive airway pressure (CPAP) or non-invasive positive airway pressure (NIPPV) devices
* Those who require long-term oxygen therapy (oxygen therapy time>15 hours/day)
* Individuals who have undergone lobectomy or lung volume reduction surgery within the 12 months prior to the start of the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) | From the use of the investigational drug until the last study visit, up to day 16
  The occurrence of all adverse events (AE) including abnormal laboratory test indicators.
Serious adverse events (SAE) | From the use of the investigational drug until the last study visit, up to day 16
  The occurrence of all serious adverse events (SAE) .
Forced expiratory volume (FEV1) trough value changed from baseline | After administration of Day1 and Day7，before administration of Day3 and Day5
  After administration of Day1 and Day7, the FEV1 trough value changed from baseline.
  The changes in FEV1 before administration of Day3 and Day5 compared to baseline.
Forced vital capacity (FVC) changes compared to baseline | After administration of Day1 and Day7，before administration of Day3 and Day5
  FVC changes compared to baseline at each lung function visit point.
The peak FEV1 value changed from baseline | After administration of Day1 and Day7，before administration of Day3 and Day5
  After administration of Day1 and Day7, the peak FEV1 value changed from baseline.
The area under the FEV1 curve of the average change from baseline | After administration of Day1 and Day7，before administration of Day3 and Day5
  The area under the FEV1 curve of the average change from baseline after administration of D1 and D7 ranges from 0-6h (AUC0-6h), 0-12h (AUC0-12h), 12-24h (AUC12-24h), 0-24h (AUC0-24h), and FVC AUC (0-24h).
The change in chronic obstructive pulmonary disease (CAT) score from baseline | After administration of Day1 and Day7，before administration of Day3 and Day5
  The change in chronic obstructive pulmonary disease (CAT) score from baseline on the day after Day7 administration.

SECONDARY OUTCOMES:
Peak concentration (Cmax) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  The Cmax is the maximum observed plasma concentration of study drug.
Area Under the Concentration-Time Curve From 0 to Last Observation (AUC [0-t]) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  To characterize the pharmacokinetics of TQC3927 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Area Under the Concentration-Time Curve From Zero to Infinity (AUC [0-infinity]) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  To characterize the pharmacokinetics of TQC3927 by assessment of area under the plasma concentration time curve from 0 extrapolated to infinity.
Time to reach maximum (peak) plasma concentration following drug administration (Tmax) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  To characterize the pharmacokinetics of TQC3927 by assessment of time to reach maximum plasma concentration after single and multiple dosing.
Half-life (t1/2) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Apparent volume of distribution(Vd/F) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  Apparent volume of distribution of the TQC3927 in plasma
Apparent clearance (CLz/F) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
End elimination rate (λz) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  Derived from semi logarithmic linear regression of eliminating phase concentration points.
Residual area percentage (AUC_%Extrap) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  Residual area percentage of the TQC3927 in plasma.
Average dwell time(MRT0-t) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  The average residence time from 0:00 to the last measurable concentration time point.
Average dwell time(MRT0-∞) | Day1: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24 hours after-dose, Day5: pre-dose, Day6: pre-dose, Day7: pre-dose, at 15,30,45 minutes,1,2,4,6,8,12,24,48,72 hours after-dose
  Average residence time from 0:00 to infinity.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - China Japan Friendship Hospital, Beijing, Beijing Municipality
  - Aerospace Center Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Heze Municipal Hospital, Heze, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - The Third People Hospital of Chengdu, Chengdu, Sichuan
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang